CLINICAL TRIAL: NCT03176719
Title: The Non-specific Effects of Vaccination Related to Mortality and Morbidity in Nanoro Health and Demographic Surveillance System Cohort
Brief Title: Non-specific Effects of Vaccination on Mortality and Morbidity
Acronym: NOVAC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Clinical Research Unit of Nanoro (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017-3339
Record Dates: First submitted 2017-05-18; First posted 2017-06-05 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Vaccine Reaction; Anemia; Malaria,Falciparum; Salmonella Bacteraemia
MeSH Terms: conditions — Anemia; Malaria, Falciparum | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — EDTA blood and heparizined blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Children of 1 years old: 200 healthy volunteers aged between 12 and 23 months
  Interventions: Other: Venipuncture
- Children aged 2-4: 200 healthy volunteers aged between 24 and 59 months
  Interventions: Other: Venipuncture
- Children aged 5 - 9: 200 healthy volunteers aged between 60 and 119 months
  Interventions: Other: Venipuncture
- Children aged 10 - 14: 200 healthy volunteers aged between 120 and 179 months
  Interventions: Other: Venipuncture
- Adults of 15 years and older: 200 healthy volunteers of 180 months or older
  Interventions: Other: Venipuncture

INTERVENTIONS:
Other: Venipuncture — 1. Full blood count and leukocyte differentiation.
  2. Detection of malaria parasites and parasite differentiation to trophozoites, gametocytes and ringstages (XN-30)
  3. Detection of anemia, thallasemia and sickle cell anemia (XN-20)
  4. Ex-vivo stimulation of wholeblood with various stimuli. Read-out will be a spectrum of cytokines (ELISA)
  5. Circulating cytokines and inflammatory markers (ELIZA)
  6. DNA analysis to assess genetic variations determining pro- versus anti inflammatory response including mTOR, HK2, PFKP, GLS, and GLUD1/2.
  7. pan-Salmonella PCR
  8. Gametocyte PCR

SUMMARY:
It has long been recognized that the positive effects of vaccination on childhood mortality cannot be solely attributed to a decline in the disease targeted by the vaccine. These so-called non-specific effects of vaccination have so far mostly been linked to mortality. However, it has been suggested that non-specific effects may also effect morbidity and nutritional status. This study aims to further explore the correlation between vaccination, susceptibility to infectious diseases (particularly malaria and bacterial infections), nutritional status and immunity.

With this prospective cross sectional study among healthy individuals in rural west-Africa we aim to address several research questions at the same time. This study will assess the influence of (time-point of) vaccination on morbidity, mortality and immune status among healthy individuals in a rural sub-Saharan African setting. Secondly, to explore the prevalence of subclinical malaria, iron deficiency anemia, sickle cell anemia and thallasemia among a healthy rural sub-Saharan African population. And finally to assess normal hemocytometry values among a healthy rural sub-Saharan African population.

DETAILED DESCRIPTION:
A cross sectional study among healthy participants randomly selected from the population living in the Nanoro HDSS cohort to (a) study the relation between vaccination and morbidity (including hemoglobin levels, subclinical malaria and stunting) (b) perform hemocytometry in order to determine reference values for that population and estimate the prevalence and causes of anemia, using reference values from other Sub-Sahara Africa countries and industrialized countries.

In a cross sectional study among a healthy population in the Nanoro HDSS cohort, hemocytometry will be performed in order to define normal values for that population. In addition, hemoglobin levels can be related to the presence of iron deficiency, thalassemia and malaria and be corrected for important confounding factors, such as the family income, family composition, distance to a healthcare center and vaccination status. This study will allow to assess simultaneously the normal range of hemoglobin values, the prevalence of (different causes of) anemia, the prevalence of subclinical malaria parasitemia, as well as the influence of (timepoint of) vaccination on all these issues. It is hypothized that early vaccination with live attenuated vaccines has a protective effect against malaria and other severe infectious diseases and will result in a better nutritional status, a higher hemoglobin level and a higher threshold of subclinical parasitemia. The protective effect of early vaccination with live attenuated vaccines may be due to the long-term modulation of the immune system through epigenetic changes causing a right balance between the pro- and anti-inflammatory responses. Such balance can be determined by ex-vivo stimulation of whole blood by a variety of stimuli, including Mycobacterium tuberculosis and lipopolysaccharide from Escherichia coli, followed by measurement of ex vivo cytokine production. Previous studies among healthy volunteers in the Netherlands have shown that BCG is indeed capable to induce epigenetic changes and influence immune response by influencing various pathways including through genetic variations in mTOR, HK2, PFKP, GLS, and GLUD1/2 (ref).

The new Sysmex analysers are not only capable to determine hemocytometry, but are at the same time capable to detect malaria parasites directly. Interestingly, not only the asexual stages of the parasites are detected but the gametocytes as well. This may be very important as gametocyte carriers are known to play a crucial role in malaria transmission. Gametocytes are presently detected by light microscopy or by PCR, however these techniques are limited; the sensitivity of light microscopy is relatively low and PCR is too complex to perform in most rural sub-Saharan African settings. The new Sysmex hematology analysers are easy to operate at low costs and may as such become an important tool for malaria elimination programs. No data are presently available about gametocyte density in Burkina Faso in a large population, nor is the lower level of detection of gametocytes using the sysmex analyzers known.

This research has four main objectives :

1. To perform hemocytometry among a healthy rural Burkina Faso population selected from the Nanoro HDSS cohort, in order to determine reference values for that population.
2. To perform hemocytometry among a healthy rural Burkina Faso population selected from the Nanoro HDSS cohort, in order to estimate the prevalence and causes of anemia, using reference values from other Sub-Sahara Africa (SSA) countries and industrialized countries.
3. To study the relation between (timepoint of) vaccination and morbidity (including hemoglobin levels, subclinical malaria, bacterial infection and stunting) among a healthy rural Burkina Faso population selected from the Nanoro HDSS cohort. For this objective the population will be stratified by birth cohort.
4. To perform ex-vivo whole blood stimulation to assess differences in immune response between patientgroups with a different vaccination status, within a healthy rural Burkina Faso population selected from the Nanoro HDSS cohort

   Seondary objectives
5. To assess the detection limit of gametocyte carriages for the new series Sysmex hematology analyzers.
6. To assess if Salmonella resides in blood as a reservoir for invasive infection among a rural Burkina Faso population selected from the Nanoro HDSS cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants currently living in the Nanoro HDSS area, born before May 2016.

Exclusion Criteria:

* Current febrile illness,
* Current chronic illnesses, HIV, TB, renal failure, cardiac disease (if known)
* Patients that have participated in the RTSS vaccination trial from Glaxo-Smith-Kline at the same inclusion site.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 5 groups will be selected. Each age group will consist of 220 participant (including 20% for potential non response). The survey will be conducted among 24 villages. Demographic age distribution is comparable for each of the villages. In order to prevent bias, a proportionate number of participants will be selected from each village based on its total population. Participants will then be randomly selected from each sample stratum using systematic selection.
Sampling Method: Non-Probability Sample
Enrollment: 1005 (Actual)
Dates: Start 2017-06-17 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Vaccination data | June 2017 - December 2017
  Vaccination data as recorded on the vaccination card
Nutritional status (Z-score or BMI) | June 2017 - December 2017
  weight (kg), height (cm) and upperarm circumference (mm) leading to outcome measure on nutritional status: as appropriate Z-score or BMI
History of disease | June 2017 - December 2017
  Recorded history of disease according to the participants health card
Immunological profile | June 2017 - December 2017
  Cytokine levels, including IL-1b, IL-6, IL-10, IFN-gamma, TNF-alpha and IL-17, which will be assessed through ELISA. Measurement will be done on stimulated and unstimulated blood. Ex-vivo whole blood stimulation will be done with RPMI, LPS, MTB, Staphylococcus aureus, Candida albicans and Salmonella Typhimurium.
Genetic immunological profile | June 2017 - December 2017
  DNA analysis to assess genetic variations determining pro- versus anti inflammatory response including mTOR, HK2, PFKP, GLS, and GLUD1/2.
subclinical parasitemia | June 2017 - December 2017
  low level malaria infection detected by SYSMEX hematology analyzer XN - 30
Anemia | June 2017 - December 2017
  Differentiation of different forms of anemia using SYSMEX hematology analyzers XN -20 and XN - 30
Reference values for hemocytometry in a healthy rural population from Burkina Faso | June 2017 - December 2017
  Hemocytometry using SYSMEX hematology analyzers XN -20 and XN - 30

SECONDARY OUTCOMES:
Gametocyte PCR | June 2017 - December 2017
  Gametocyte PCR on EDTA whole blood stored in RNA protect

OTHER OUTCOMES:
Salmonella PCR | June 2017 - December 2017
  Salmonella PCR on EDTA whole blood (ethical clearance not yet obtained, amendment in progress)

CONTACTS AND LOCATIONS:
Overall Officials: André van der Ven, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Clinical Research Unit of Nanoro, Nanoro, Boulkiemedé, Burkina Faso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kabore B, Post A, Berendsen MLT, Diallo S, Lompo P, Derra K, Rouamba E, Jacobs J, Tinto H, de Mast Q, van der Ven AJ. Red blood cell homeostasis in children and adults with and without asymptomatic malaria infection in Burkina Faso. PLoS One. 2020 Nov 30;15(11):e0242507. doi: 10.1371/journal.pone.0242507. eCollection 2020. PMID 33253198